CLINICAL TRIAL: NCT05131555
Title: Influence of Endurance Training and Histamine Receptor Antagonists on the Transcriptome Response in Human Muscle
Brief Title: Influence of Endurance Exercise and Histamine Receptors on the Gene Expression in Skeletal Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: AET - BC-10237
Record Dates: First submitted 2021-10-15; First posted 2021-11-23 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Exercise; Histamine
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded placebo-controlled cross-over interventional study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1: Placebo (Placebo Comparator): lactose
  Interventions: Drug: Placebo: Placebo + exercise training.
- H1 blockade (Experimental): 540 mg Fexofenadine
  Interventions: Drug: H1 blockade: H1 receptor antagonist + exercise training
- H2 blockade (Experimental): 40 mg Famotidine
  Interventions: Drug: H2 Blockade: H2 receptor antagonist + exercise training

INTERVENTIONS:
Drug: Placebo: Placebo + exercise training. — Oral placebo Exercise training: Interval-based cycling exercise
  Arms: 1: Placebo
Drug: H1 blockade: H1 receptor antagonist + exercise training — H1 blockade: oral blockade Exercise training: Interval-based cycling exercise
  Arms: H1 blockade
Drug: H2 Blockade: H2 receptor antagonist + exercise training — H2 blockade: oral blockade Exercise training: Interval-based cycling exercise
  Arms: H2 blockade

SUMMARY:
Blocking histamine H1/H2 receptors blunts chronic endurance training adaptations. The current study addresses a twofold research question: "What is the influence of endurance training (1) and histamine H1 and H2 signaling (2) on the gene expression in human skeletal muscle." Results from this study will yield more insights into the molecular mechanisms of adaptations to exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* 18-45 years
* not to medium physically active

Exclusion Criteria:

* Smoking
* Chronic disease
* Supplement or medication intake
* Seasonal allergies

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in muscle transcriptome (direct response) | On each test-day: 0 minutes after the exercise training versus at rest.
  RNA-sequencing
Change in muscle transcriptome (delayed response) | On each test-day: 180 minutes after the exercise training versus at rest.
  RNA-sequencing
Muscle glycogen depletion | On each test-day: 0 minutes after the exercise training versus at rest.
  Fluorometric determination of muscle glycogen levels
Muscle glycogen resynthesis | On each test-day: 180 minutes after the exercise training versus at rest.
  Fluorometric determination of muscle glycogen levels
Plasma volume change | Change from rest to different time-points after exercise (0, 30, 60, 120 and 180 minutes after the exercise training).
  Plasma volume based on hemoglobin and hematocrit concentration.

SECONDARY OUTCOMES:
Heart rate during the exercise training | Continuously during training on each test-day.
  Heart rate during the exercise training.
Blood lactate | On each test-day at 10 time-points: at rest, during exercise and 0, 30, 60, 120 and 180 minutes after the exercise training.
  Capillary lactate concentration.
Blood glucose | On each test-day at 10 time-points: at rest, during exercise and 0, 30, 60, 120 and 180 minutes after the exercise training.
  Capillary glucose concentration.
Blood histamine | On each test-day at 6 time-points: at rest and 0, 30, 60, 120 and 180 minutes after the exercise training.
  histamine concentration in blood samples.
Blood insulin | On each test-day at 6 time-points: at rest and 0, 30, 60, 120 and 180 minutes after the exercise training.
  insulin concentration in blood samples.
Muscle signaling pathways relevant for glucose metabolism and cardiovascular health | On each test-day: at rest, 0 minutes and 180 minutes after the exercise training.
  Phosphorylation status of proteins assessed by Western Blotting

CONTACTS AND LOCATIONS:
Overall Officials: Wim Derave, Professor, Principal Investigator — University Ghent
Locations (1):
- Department of movement and sports sciences, Ghent University, Belgium, Ghent, Oost-Vlaanderen, Belgium